CLINICAL TRIAL: NCT01426360
Title: A Randomized, Double-blind Clinical Trial to Assess the Instant and Lasting Relief Effects of a Dentifrice Containing 2% Strontium Chloride and 5% Potassium Nitrate on Dentin Hypersensitivity
Brief Title: Instant and Lasting Relief Effects of Strontium Chloride/Potassium Nitrate Dentifrice on Dentin Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Liu Hongchun, Ph.D, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DH-38
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Results first posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-11

CONDITIONS: Dentine Hypersensitivity
Keywords: dentifrice; potassium nitrate; strontium chloride
MeSH Terms: conditions — Dentin Sensitivity | interventions — strontium chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- strontium chloride/potassium nitrate dentifrice (Experimental)
  Interventions: Other: strontium chloride/potassium nitrate dentifrice
- control dentifrice (Placebo Comparator)
  Interventions: Other: control dentifrice

INTERVENTIONS:
Other: control dentifrice — use the dentifrice to brush teeth twice a day for one minute for 3 days
  Arms: control dentifrice
Other: strontium chloride/potassium nitrate dentifrice — use the dentifrice to brush teeth twice daily for 3 days
  Arms: strontium chloride/potassium nitrate dentifrice

SUMMARY:
The objective of the present study was to compare the effects of a commercially available dentifrice containing 2% strontium chloride and 5% potassium nitrate in a silica base, versus a control dentifrice, containing exactly the same ingredients apart from strontium chloride and potassium nitrate, on the instant and lasting relief of DH.

DETAILED DESCRIPTION:
Dentin hypersensitivity (DH) is a very common complaint that occurs in the general population. The intensity of the pain can be minor to very serious, which may prevent one from eating or performing ordinary oral hygiene practices. The most accepted mechanism by which DH occurs is hydrodynamic theory, which suggests that pain-producing stimuli cause rapid movement of fluid within the dentin tubules, as a result the free nerve endings, at the inner ends of the tubules or the periphery of the pulp, are excited and DH occurs. According to this theory, one approach to treat DH is reducing dentin tubule fluid movement through occluding open tubules. Strontium chloride was the first tubule-blocking ingredient used in dentifrice about fifty years ago and since that time a paucity of clinical studies have been carried out to test its effectiveness on DH. The other approach is to reduce the pulp nerve excitability by depolarizing the nerve endings, in which the most widely used material is potassium salts. Although there is limited clinical evidence that dentifrices containing strontium chloride or potassium nitrate alone, as the major desensitizing agent, has an effect on reducing DH, no clinical studies have shown the effectiveness of a dentifrice containing both strontium chloride and potassium nitrate in a silica base on alleviating DH.

ELIGIBILITY:
Inclusion Criteria:

* good oral and general health
* possessing at least two teeth (incisors, cuspids, bicuspids and first molars with exposed cervical dentin) with hypersensitivity on facial surfaces which satisfied a tactile hypersensitivity stimulus score of 10-50 grams of force (Yeaple probe) and an air blast stimulus score of 2 or 3(Schiff Cold Air Scale)
* provided informed consent and were available for the study duration

Exclusion Criteria:

* progressive periodontitis, with teeth that had extensive restoration, suspected pulpitis, caries, cracked enamel or that were used as abutments for removable partial dentures,
* had hypersensitive teeth with a mobility greater than one
* had received periodontal treatment including surgery during the last year
* had used any other anti-hypersensitivity dentifrice or taken part in any other clinical trial, used any desensitizing agents during the last three months, or allergic to the ingredients of the dentifrices were excluded
* pregnant or breastfeeding women
* had taken the following drugs during the last month: anticonvulsants, antihistamines, antidepressants, sedatives, tranquilizers, anti-inflammatory drugs or daily analgesics

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hongchun Liu, Ph.D., Principal Investigator — Department of Preventive Dentistry,Guanghua College of Stomatology,Sun Yat-sen University
Locations (1):
- the State Key Laboratory of Oral Diseases, Sichuan University, Chengdu, China, Chengdu, Sichuan, China

REFERENCES:
- [Background] Fu Y, Li X, Que K, Wang M, Hu D, Mateo LR, DeVizio W, Zhang YP. Instant dentin hypersensitivity relief of a new desensitizing dentifrice containing 8.0% arginine, a high cleaning calcium carbonate system and 1450 ppm fluoride: a 3-day clinical study in Chengdu, China. Am J Dent. 2010 May;23 Spec No A:20A-27A. PMID 21284248
- [Derived] Liu H, Hu D. Efficacy of a commercial dentifrice containing 2% strontium chloride and 5% potassium nitrate for dentin hypersensitivity: a 3-day clinical study in adults in China. Clin Ther. 2012 Mar;34(3):614-22. doi: 10.1016/j.clinthera.2012.01.027. Epub 2012 Mar 3. PMID 22385928

RESULTS

PARTICIPANT FLOW:
Groups:
- Strontium Chloride/Potassium Nitrate Dentifrice: Subjects receive a commercially available dentifrice containing 2% strontium chloride and 5% potassium nitrate in a silica base (the experimental group)
- Control Dentifrice: Subjects receive a commercially available control dentifrice containing exactly the same ingredients with the exception of strontium chloride and potassium nitrate (the control group)
Period: Overall Study
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Started | 38 | 41
Completed | 38 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 38 | 41 | 79
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.37 (8.8) | 43.39 (8.8) | 42.9 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 55
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  China | 38 | 41 | 79
Baseline tactile hypersensitivity score [Mean (Standard Deviation); unit: gram] — Tactile hypersensitivity assessments were done using an Electronic Force Sensing Probe (Yeaple Probe Model 200A, Xinix Research Inc., USA). Scores were recorded in terms of a quantified, reproducible force applied by a #19 explorer tip. After presetting the probe to 10 grams, the tip of the probe was run across the exposed dentin perpendicular to the examined surface. Subsequent passes were made, each time the applied force was increased by 10 grams, until the subject indicated that he/she was experiencing discomfort, or until the maximum force of 50 grams had been reached.
  gram | 12.63 (5.16) | 12.2 (3.72) | 12.41 (4.45)
Baseline air blast hypersensitivity score [Mean (Standard Deviation); unit: Scores on a scale] — The tooth was isolated. Air was delivered from a standard dental unit air syringe and directed at the exposed buccal surface of the hypersensitive tooth for 1 second. The Schiff Cold Air Sensitivity Scale was used to assess the subjects' response.
  0 - Subject does not respond to air stimulus;
  1. - Subject responds to air stimulus, but does not request discontinuation of stimulus;
  2. - Subject responds to air stimulus and requests discontinuation or moves from stimulus;
  3. - Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
  Scores on a scale | 2.42 (0.41) | 2.46 (0.41) | 2.44 (0.41)

OUTCOME MEASURES:

1. Primary Outcome: Tactile Hypersensitivity Scores Immediately After Topical Dentifrice Use
Description: Immediately after dentifice use, tactile hypersensitivity assessments were done using an Electronic Force Sensing Probe (Yeaple Probe Model 200A, Xinix Research Inc., USA). Scores were recorded in terms of a quantified force applied by a #19 explorer tip. After presetting the probe to 10 grams, the tip of the probe was run across the exposed dentin perpendicular to the examined surface. Subsequent passes were made, each time the applied force was increased by 10 grams, until the subject indicated that he/she was experiencing discomfort, or until the maximum force of 50 grams had been reached.
Time Frame: immediately after dentifrice use
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Number analyzed (Participants) | 38 | 41
gram | 19.47 (14.69) | 14.27 (5.76)

2. Primary Outcome: Air Blast Hypersensitivity Scores Immediately After Topical Dentifrice Use
Description: The tooth was isolated. Air was delivered from a standard dental unit air syringe and directed at the exposed buccal surface of the hypersensitive tooth for 1 second. The Schiff Cold Air Sensitivity Scale was used to assess the subjects' response.
  0 - Subject does not respond to air stimulus;
  1. - Subject responds to air stimulus, but does not request discontinuation of stimulus;
  2. - Subject responds to air stimulus and requests discontinuation or moves from stimulus;
  3. - Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Time Frame: immediately after dentifrice use
Measure: Mean (Standard Deviation); unit: scale
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Number analyzed (Participants) | 38 | 41
scale | 1.93 (0.51) | 2.22 (0.6)

3. Primary Outcome: Tactile Hypersensitivity Score After 3 Days of Dentifrice Use
Description: After 3 days, tactile hypersensitivity assessments were done using an Electronic Force Sensing Probe (Yeaple Probe Model 200A, Xinix Research Inc., USA). Scores were recorded in terms of a quantified, reproducible force applied by a #19 explorer tip. After presetting the probe to 10 grams, the tip of the probe was run across the exposed dentin perpendicular to the examined surface. Subsequent passes were made, each time the applied force was increased by 10 grams, until the subject indicated that he/she was experiencing discomfort, or until the maximum force of 50 grams had been reached.
Time Frame: 3 days after dentifrice use
Measure: Mean (Standard Deviation); unit: gram
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Number analyzed (Participants) | 38 | 41
gram | 19.87 (14.95) | 14.27 (5.98)

4. Primary Outcome: Air Blast Hypersensitivity Score 3 Days After Dentifrice Use
Description: After 3 days, tooth was isolated. Air was delivered from a standard dental unit air syringe and directed at exposed buccal surface of the hypersensitive tooth for 1 second. The Schiff Cold Air Sensitivity Scale was used to assess the subjects' response.
  0 - Subject does not respond to air stimulus;
  1. - Subject responds to air stimulus, but does not request discontinuation of stimulus;
  2. - Subject responds to air stimulus and requests discontinuation or moves from stimulus;
  3. - Subject responds to air stimulus, considers stimulus to be painful, and requests discontinuation of the stimulus.
Time Frame: 3 days after dentifrice use
Measure: Mean (Standard Deviation); unit: scale
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Number analyzed (Participants) | 38 | 41
scale | 1.8 (0.56) | 2.13 (0.6)

ADVERSE EVENTS:
Arm/Group | Strontium Chloride/Potassium Nitrate Dentifrice | Control Dentifrice
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/38 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No